CLINICAL TRIAL: NCT05629663
Title: Utilizing of Augmented Reality Technology for Development, Application and Evaluation on Nurse Education Program
Brief Title: Utilizing of Augmented Reality Technology Education Program for Nurse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-08-079
Record Dates: First submitted 2022-10-10; First posted 2022-11-29 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2022-10

CONDITIONS: Nursing; Education
Keywords: Nursing; Education; Augmented reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AR program group (Experimental): participants in the AR group were guided by AR-based instructions and requested assistance with the head-mounted device.
  Interventions: Device: AR guidance with Hololens 2

INTERVENTIONS:
Device: AR guidance with Hololens 2 — The AR instructions were developed as a step-by-step guide, utilizing the dynamic 365 Guide (Software, Microsoft Corporation, Redmond, WA, USA). The AR instructions were delivered using the Microsoft HoloLens 2.

SUMMARY:
It is important to provide practice-oriented education for nurses in a safe environment. As it became difficult to maintain face-to-face education and practice environment due to COVID-19, a new paradigm for nurse education was required. The investigators tried to use augmented reality technology in nurse education, and based on this, research was conducted to devise, develop, apply, and evaluate the satisfaction and usability of educators. The field needs were checked through literature review, the subject of the augmented technology-based education program was selected, and the program was produced and applied, and this was evaluated through a questionnaire including a system usability evaluation scale and a technology acceptance model-based question.

DETAILED DESCRIPTION:
As patient-centered nursing education is considered more important, the amount of nursing education required is also increasing. In addition, the safety of the educational environment is important for nurses' application education to various clinical environments. In the past, simulation education, which generally expects learning effects through practice and motivation, was mainly conducted. However, in the COVID-19 situation, it has become difficult for educators and educators to gather in one space to conduct clinical education.[4] Based on the need for alternatives to this, The investigators devised a nurse education program using various new technologies.

Recently, virtual training systems are being developed in various application fields thanks to the development of augmented reality and virtual reality. In particular, medical training and clinical application have become important since the recent international epidemic of COVID-19. The strength of new technologies such as Augmented Reality (AR) has enabled various programs for education and healthcare that have overcome the limitations of time and space. Augmented reality is already being applied to self-directed learning in various areas, which provides learners with a highly immersive learning environment so that medical personnel can receive more accurate and precise medical education in the field.

The investigators tried to develop an augmented reality technology-based program that can provide training to nurses using the Headmount display device, and to find out the evaluation that reaches usability and satisfaction after applying it to educators.

ELIGIBILITY:
Inclusion Criteria:

* Medical staff who have participated, trained or trained in the production of ventilator/ECMO training programs using HoloLens 2
* A person who has agreed to voluntarily participate in the study through the recruitment notice

Exclusion Criteria:

* Medical staff who participate, train, or have not been trained in the production of ventilator/emo education programs using HoloLens 2
* Medical staff who participated, trained, uneducated, or abandoned in the production of ventilator/emo education programs using HoloLens 2 If you disagree with the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Device Usability and Feasibility Evaluation | day1
  Semi-structured interviews will be conducted to evaluate the feasibility and usability of the device. The interview will focus on user experiences, operational feasibility, and feedback on device design and functionality. The questions will assess ease of use, clarity of instructions, and perceived benefits.

SECONDARY OUTCOMES:
System usability scale | day1
  survey for System Usability Scale. a five-point scale(1 point to 5 point), High scores can be positive for each question, and low scores can be positive.
Technology acceptance scale | day1
  It consists of 15 questions that assess trends in the latest technology with questions on a scale of 1 to 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Centre, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoo S, Heo S, Song S, Park A, Cho H, Kim Y, Cha WC, Kim K, Son MH. Adoption of Augmented Reality in Educational Programs for Nurses in Intensive Care Units of Tertiary Academic Hospitals: Mixed Methods Study. JMIR Serious Games. 2024 May 23;12:e54188. doi: 10.2196/54188. PMID 38780998